CLINICAL TRIAL: NCT05179070
Title: The Effect of Carvedilol Rapid Up-Titration in Patients With Heart Failure With Reduced Ejection Fraction (Biomolecular and Clinical Study on IL-6, TNF-α, NT-ProBNP, MDA, LVEF, 6MWT, and KCCQ)
Brief Title: Effect of Carvedilol Rapid Up-Titration in Patients With Heart Failure With Reduced Ejection Fraction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, dr. Habibie Arifianto Sp.JP(K)., M.Kes., FIHA, Principal Investigator, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001/02/08/90
Record Dates: First submitted 2021-11-17; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction HFrEF
Keywords: HFrEF; Carvedilol; Rapid UpTitration; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: Devided into 2 groups. The first is the rapid up-titration group, which will get carvedilol up-titration every day, 3.125mg twice daily on the first day, 6.125mg twice daily on the second day, 12.5mg twice daily on the third day and 25mg twice daily on the fourth day consecutively. And the second group will have carvedilol titration according to established guidelines on Heart Failure, start 3.125mg twice daily, and up titrated every 2 weeks
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient, Care Provider and Investigator didn't know about dose of carvedilol and grouping of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UpTitration (Experimental): the first is the rapid up-titration group, which will get carvedilol up-titration every day, 3.125mg twice daily on the first day, 6.125mg twice daily on the second day, 12.5mg twice daily on the third day and 25mg twice daily on the fourth day consecutively
  Interventions: Drug: Carvedilol
- Control (Active Comparator): And the second group will have carvedilol titration according to established guidelines on Heart Failure, start 3.125mg twice daily, and up titrated every 2 weeks
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — the first is the rapid up-titration group, which will get carvedilol up-titration every day, 3.125mg twice daily on the first day, 6.125mg twice daily on the second day, 12.5mg twice daily on the third day and 25mg twice daily on the fourth day consecutively. And the second group will have carvedilol titration according to established guidelines on Heart Failure, start 3.125mg twice daily, and up titrated every 2 weeks
  Other Names: Vblock

SUMMARY:
Guidelines-directed medical therapy has improved dramatically outcomes in heart failure with reduced ejection fraction (HFrEF) patients. Beta-blockers have the most beneficial effects on all caused mortality and rehospitalization on HFrEF, but unfortunately, since the discovery of beta-blocker therapy in HFrEF, there was no change in the way of titration, start low go slow, which resulted in difficulties in reaching optimal doses for some patients.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, single-center study in HFrEF patients, that held in Universitas Sebelas Maret Hospital, Central Java, Indonesia. The investigators divided 26 HFrEF patients consecutively into two groups, the first is the rapid up-titration group, which will get carvedilol up-titration every day, 3.125mg twice daily on the first day, 6.125mg twice daily on the second day, 12.5mg twice daily on the third day and 25mg twice daily on the fourth day consecutively. And the second group will have carvedilol titration according to established guidelines on Heart Failure, start 3.125mg twice daily, and up titrated every 2 weeks. Every patient will be checked for IL-6, TNF-α, NT-ProBNP, MDA, left ventricular Ejection Fraction, six minutes walking test, and Kansas City Cardiomyopathy Questionnaire on day 1, pre-discharge, and one month after hospitalization. The study was approved by the university ethics committee. The clinical parameters evaluated at admission were analyzed using variable comparative with Shapiro Wilk or one-way ANOVA, with three intervals analysis using repeated ANOVA (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Acute heart failure patient with reduced ejection fraction in Universitas Sebelas Maret Hospital with naive betablocker therapy
* Age >18 years old
* Initial Heart Rate > 50 bpm

Exclusion Criteria:

* Cardiogenic Shock
* Septicaemia
* High degree AV Block or on pace maker
* History of beta blocker intolerance
* Reactive Pulmonary disease
* Severe Peripheral artery disease
* Creatinine level > 2.5 mg/dl
* Potassium serum >5 mmol/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Improvements of Biomolecular Parameters | 1 month
  IL-6 in pg/ml, TNF-α in pg/ml, NT-ProBNP in pg/ml, Malondyaldehide nmol/ml
Improvements of Clinical Parameters | 1 month
  Kansas City Cardiomyopathy Questionnaire (KCCQ) scores are scaled 0-100 (the higher score indicates a better condition) and 6 Minutes Walking Test in meters
Improvements of Echocardiography Parameters | 1 month
  LVEF

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 1 month
  All cause cardiac rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Habibie Arifianto, MD, Principal Investigator — Universitas Sebelas Maret
Locations (1):
- Universitas Sebelas Maret Hospital, Sukoharjo, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
This study purpose is to obtain a doctoral degree, there was no sponsorship during this study therefore the IPD cannot be shared

REFERENCES:
- [Background] Wolfe NK, Mitchell JD, Brown DL. The independent reduction in mortality associated with guideline-directed medical therapy in patients with coronary artery disease and heart failure with reduced ejection fraction. Eur Heart J Qual Care Clin Outcomes. 2021 Jul 21;7(4):416-421. doi: 10.1093/ehjqcco/qcaa032. PMID 32324852
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Am Coll Cardiol. 2017 Aug 8;70(6):776-803. doi: 10.1016/j.jacc.2017.04.025. Epub 2017 Apr 28. No abstract available. PMID 28461007
- [Background] Martinez-Selles M, Datino T, Alhama M, Barrueco N, Castillo I, Fernandez-Aviles F. Rapid carvedilol up-titration in hospitalized patients with left ventricular systolic dysfunction--data from the Carvedilol in Hospital: Up-titration Limits after Acute Patients Admission registry. J Cardiovasc Med (Hagerstown). 2010 May;11(5):352-8. doi: 10.2459/JCM.0b013e328334f48b. PMID 20154635
- [Result] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191